CLINICAL TRIAL: NCT07208136
Title: An Open-label, Multi-center Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of JMKX005425 Tablets in Subjects With Microsatellite Instability-High or Mismatch Repair Deficient Advanced Solid Tumors
Brief Title: A Study of JMKX005425 in Patients With MSI-H/dMMR Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMKX005425-X101
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JMKX005425 (Experimental): Subjects will take a pre-specified dose of JMKX005425.
  Interventions: Drug: JMKX005425

INTERVENTIONS:
Drug: JMKX005425 — JMKX005425 administered orally.

SUMMARY:
This is a first-in-human, Phase I, open-label, multi-center, dose-escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of JMKX005425 in subjects with microsatellite instability-high (MSI) and/or mismatch repair deficiency (dMMR) advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have a microsatellite instability-high (MSI) and/or mismatch repair deficiency (dMMR), histologically or cytologically documented advanced solid tumor.
2. Has at least one measurable lesion per RECIST v1.1.
3. Has a life expectancy of ≥ 12 weeks.
4. Adequate organ function.

Exclusion Criteria:

1. Toxicities from prior anti-tumor therapy has not recovered to Grade 1 or below per CTCAE v5.0.
2. History of prior malignancy in the past 3 years, with the exception of curatively treated malignancies.
3. Has the dysphagia, or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drug.
4. Has the severe chronic or active infection
5. Has a history of severe cardiovascular disease.
6. Subject is pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs), AEs, serious AEs (SAEs) | up to 2 years
  To assess the safety and tolerability of JMKX005425.

SECONDARY OUTCOMES:
maximum plasma concentration (Cmax) | Up to 2 months
  Maximum observed concentration.
maximum plasma concentration (Tmax) | Up to 2 months
  Time to reach maximum observed plasma concentration.
Objective Response Rate (ORR) | Up to 2 years
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease Control Rate (DCR) | Up to 2 years
  DCR is the percentage of patients with a best overall response of CR or PR or Stable Disease (SD) per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China